CLINICAL TRIAL: NCT04970784
Title: Impact of a Dedicated Geriatric Sector on the Loss of Functional Autonomy at 1 Month for Patients Admitted to Emergencies and Non-hospitalised
Acronym: URG-GERIA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0973; 2020-A00211-38 (Other: ID-RCB)
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Health Services for the Aged; Emergency Service, Hospital; Ambulatory Care
Keywords: Elderly; Geriatric sector; Autonomy
MeSH Terms: conditions — Emergencies | interventions — Activities of Daily Living; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients cared for by the adult sector: Patients admitted to emergencies, non-hospitalized and cared for by the adult sector of emergencies (classical emergencies)
  Interventions: Other: Activities of Daily Living (ADL) questionnaire (The Katz index )
- Patients cared for by the geriatric sector: Patients admitted to emergencies, non-hospitalized and cared for by the geriatric sector of emergencies
  Interventions: Other: Activities of Daily Living (ADL) questionnaire (The Katz index )

INTERVENTIONS:
Other: Activities of Daily Living (ADL) questionnaire (The Katz index ) — For patients cared for by the geriatric sector, questionnaire will be filled in at admission D0 and by phone at D30, for the "classic" emergency patients questionnaire will be submitted by phone the day following the consultation D1, and D30.

SUMMARY:
Several studies have shown that going to the emergency room is a risk factor for loss of independence in the elderly. It has been shown that the period following an emergency room visit without hospitalization is a period of vulnerability for the elderly.

The functional decline, or loss of functional autonomy, of the elderly is associated with an increase in institutionalization, mortality and costs to society.

Studies have highlighted the risk factors for functional decline in the elderly, such as pre-existing functional and cognitive decline, undernutrition, but no model of care has yet prevented the risk of loss of autonomy after a stay in the emergency room.

A full and early geriatric assessment could prevent functional decline after the emergency room visit.

The primary objective of the study is to assess the impact of a dedicated geriatric sector on the functional decline at 1 month of patients admitted to emergencies without hospitalization by comparing an intervention group (patient having benefited from the geriatric sector) and a group witness ("classic" emergency patient).

The secondary objective is to evaluate the impact of this sector on the number of falls at home as well as the readmission rate within 1 month of going to the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 75 years
* Emergency room consultation between 7:30 a.m. and 5:30 p.m.
* Relevant to the adult emergency department
* Return home after consultation

Exclusion Criteria:

* Age less than 75 years
* Arrival time between 5.30 p.m. and 7.30 a.m.
* Need to take care of unhooking
* Belonging to the short sector, versatile sector
* Patients hospitalized after consultation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients admitted to emergencies without hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Change of functional decline at 1 month, measured by the Katz index, Activities of Daily Living (ADL) | At Baseline (admission to ermergencies) and 1 month
  The Katz index, Activities of Daily Living (ADL) questionnaire, assess through 6 items (ranging from 0 to 1) the aptitude to execute daily life activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica POINTURIER, Principal Investigator — Centre Hospitalier Alpes Léman, service des urgences
Locations (1):
- Centre Hospitalier Alpes Léman, service des urgences, Contamine-sur-Arve, France